CLINICAL TRIAL: NCT06526403
Title: Echocardiography-Guided Percutaneous Closure of Oval-Shaped Secundum Atrial Septal Defects
Brief Title: Echocardiography-guided Oval-shaped ASD Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB.02.01/VII/020/KEP020/2023
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: ASD II; Percutaneous Closure; Zero-fluoroscopy

STUDY DESIGN:
Intervention Model Description: Zero-fluoroscopy oval-shaped secundum ASD closure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zero fluoroscopy oval-shaped secundum ASD closure (Experimental)
  Interventions: Device: Zero-fluoroscopy ASD closure

INTERVENTIONS:
Device: Zero-fluoroscopy ASD closure — Percutaneous ASD closure without fluoroscopy was performed in secundum-type oval-shaped ASD

SUMMARY:
Background: An atrial septal defect (ASD) is considered oval-shaped when its shortest diameter is less than 75% of its longest diameter. Research on the percutaneous closure of oval-shaped ASDs is limited, and to our knowledge, there are no reports of non-fluoroscopic closure for this specific population.

Objective: To assess the effectiveness of non-fluoroscopic percutaneous closure for oval-shaped ASDs.

Methods: This single-center, retrospective study examines patients undergoing percutaneous closure of oval-shaped ASDs using a non-fluoroscopy technique for initial decision-making. The device was selected to be approximately 0-4 mm larger than the longest diameter of the defect, based on measurements from transthoracic and transesophageal ultrasound.

DETAILED DESCRIPTION:
Background: An atrial septal defect (ASD) is considered oval-shaped when its shortest diameter is less than 75% of its longest diameter. Research on the percutaneous closure of oval-shaped ASDs is limited, and to our knowledge, there are no reports of non-fluoroscopic closure for this specific population.

Objective: To assess the effectiveness of non-fluoroscopic percutaneous closure for oval-shaped ASDs.

Methods: This single-center, retrospective study examines patients undergoing percutaneous closure of oval-shaped ASDs using a non-fluoroscopy technique for initial decision-making. The device was selected to be approximately 0-4 mm larger than the longest diameter of the defect, based on measurements from transthoracic and transesophageal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Oval-shaped secundum ASD with evidence of right ventricular overload, no significant and irreversible pulmonary arterial hypertension, no significant arrhythmia, no serious problems in other organs, and presumption of appropriate rims for device implantation

Exclusion Criteria:

* Other than stated in inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-07-14 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Success rate | five years

CONTACTS AND LOCATIONS:
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided